CLINICAL TRIAL: NCT05849701
Title: Shock Wave Versus Vacuum-assisted Closure on Chronic Diabetic Foot Ulcer
Brief Title: Shock Wave Versus Vacuum Assisted Closure on Chronic Diabetic Foot Ulcer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Shaimaa Mohamed Ahmed Elsayeh, Lecturer of physical therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T/INTG/3/2023/45
Record Dates: First submitted 2023-04-24; First posted 2023-05-09 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Chronic Diabetic Foot Ulcer
Keywords: Shock wave therapy; vacuum-assisted closure; Chronic diabetic foot ulcer
MeSH Terms: interventions — Extracorporeal Shockwave Therapy; Negative-Pressure Wound Therapy

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shock wave therapy group (Active Comparator): Patients in this group were managed by shock wave therapy, using gymna Shock Master 500 with an input voltage of alternating current (AC) 220 Volte, 100 pulses at 0.13 m joule/mm at 3 Hz per session, for six weeks
  Interventions: Device: Shock wave therapy
- Vacuum-assisted closure group (Active Comparator): the patients in this group were treated by vacuum-assisted closure using KCI's Vacuum Assisted Closure Device, the pump delivered an intermittent negative pressure of -125 mmHg. The cycle was of seven minutes during which the pump was on for five minutes and off for two minutes, The dressings were changed on the fourth day.
  Interventions: Device: Vacuum-assisted closure

INTERVENTIONS:
Device: Shock wave therapy — using gymna Shock Master 500 with an input voltage of alternating current (AC) 220 Volte, 100 pulses at 0.13 m joule/mm at 3 Hz per session for 6 weeks.
  Other Names: Traditional medical and wound care
  Arms: Shock wave therapy group
Device: Vacuum-assisted closure — Using KCI's Vacuum Assisted Closure Device for six weeks, the pump delivered an intermittent negative pressure of -125 mmHg. The cycle was of seven minutes during which the pump was on for five minutes and off for two minutes, the dressings were changed on the fourth day.
  Other Names: Traditional medical and wound care
  Arms: Vacuum-assisted closure group

SUMMARY:
This study will be a randomized, open-label, pretest post-test with two study groups.

DETAILED DESCRIPTION:
The randomization procedure will be performed by a simple drawing of lots (A or B) which determined whether participants would receive Shock wave therapy ( group A) or vacuum-assisted closure therapy (group B). Patients in both groups will receive the same medical treatment and nursing care.

ELIGIBILITY:
Inclusion Criteria:

All patients had chronic diabetic foot ulcers that did not heal within six weeks of the incidence.

Exclusion Criteria:

Patients with acute cellulitis, osteomyelitis, or gangrene anywhere in the affected extremity.

Patients with renal, hepatic, neurological, or malignant diseases.

Patients with severe protein malnutrition (serum albumin < 2.0 g/dl) or severe anemia (Hgb < 7.0 g/dl).

Patients with an ankle-brachial index < 0.7, absence of the dorsalis pedis or posterior tibial artery pulse.

Patients who had debridement; pregnancy.

Patients who refused to join the study, or to sign the written consent.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2023-02-14 (Actual); Study Completion 2023-04-15 (Actual)

PRIMARY OUTCOMES:
Wound surface area | change from baseline and after six weeks of intervention.
  using the ruler method to to measure the longest length and the widest width and multiplying them.
Wound volume | change from baseline and after six weeks of intervention.
  using the ruler method to to measure the longest length, the widest width and the deepest area multiplying them.

SECONDARY OUTCOMES:
Wound surface area | change from baseline and after two weeks of intervention.
  using the ruler method to to measure the longest length and the widest width and multiplying them.
Wound surface area | change from baseline and after four weeks of intervention.
  using the ruler method to to measure the longest length and the widest width and multiplying them.
Wound volume | change from baseline and after two weeks of intervention.
  using the ruler method to to measure the longest length, the widest width and the deepest area multiplying them.
Wound volume | change from baseline and after four weeks of intervention.
  using the ruler method to to measure the longest length, the widest width and the deepest area multiplying them.

CONTACTS AND LOCATIONS:
Overall Officials: Shaimaa MA El Sayeh, PhD, Principal Investigator — Lecturer at Faculty of Physical Therapy, Cairo University; Nesrein A Abdel Rashed, PhD, Principal Investigator — Assistant Professor at Faculty of Physical Therapy, Cairo University; Hamada A Hamada, PhD, Principal Investigator — Assistant Professor at Faculty of Physical Therapy, Cairo University
Locations (1):
- Shaimaa Mohamed Ahmed El Sayeh, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No